CLINICAL TRIAL: NCT07401355
Title: Improved Management of Soft Tissue Sarcomas Patients With an Optimized and Innovative Sorting Technology for Circulating Tumor Cells
Acronym: LIGHT-CTC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ET25-243 (LIGHT-CTC)
Record Dates: First submitted 2026-01-12; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Diagnosis of Soft Tissue Sarcoma (STS)
Keywords: Oncology; Soft tissue sarcoma; CTC
MeSH Terms: conditions — Neoplasms; Sarcoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- clinico-biological cohort (Other): A clinico-biological cohort with collection of tumor and blood sample for detecting and sorting circulating tumor cells
  Interventions: Other: Collection of tumor and blood sample

INTERVENTIONS:
Other: Collection of tumor and blood sample — Collection of tumor and blood sample for detecting and sorting circulating tumor cells

SUMMARY:
This trial is a monocentric, clinico-biological cohort study with prospective enrollment, aiming to develop a method for detecting and sorting CTCs (circulating tumour cells) from liquid biopsies (fresh blood samples) in patients with advanced or metastatic soft tissue sarcomas.This study include collection of clinical data, of tumor samples (collected during standard of care).

DETAILED DESCRIPTION:
EXPERIMENTAL PLAN One archival tumor sample (any FFPE and/or frozen tumor sample from surgery specimen or biopsy) will be collected.

1. A supplementary blood sample (2*10 mL EDTA) will be also collected: blood sample will be collected before anthracyclin treatment initiation and during a standart sample performed after validation of inclusion.
2. Biological analyses will be initiated once inclusion has been confirmed (See Section 6.4)
3. A supplementary blood sample (2*10 mL EDTA) will be also collected: blood sample will be collected before each chemotherapy administration and during a standart sample.
4. A supplementary blood sample (2*10 mL EDTA) will be also collected: blood sample will be collected at each disease progression and during a standart sample.
5. In case of disease progression and if a biopsy is required for the management of the patient, a tumor sample will be collected (if patient agreed and if pathological material is the sufficient).
6. Clinical data will be collected into the study eCRF. Medical FU include visits at each chemotheapy administration, and disease assessment

A total of 100 patients will be enrolled.

Considering the nature of this trial, the sample size was defined in an empirical manner considering that over the 36-month enrollment period, 100 patients could be enrolled.

The percentage of patients with detectable CTC (primary criterion) will be given with its associateed 95% confidence interval. For the seondary criteria, qualitative variables will be described using frequency and percentage distributions. The number of missing data will be given, but will not be considered for the calculation of proportions. Quantitative data will be described using the number of observations, mean, standard deviation, median, minimum and maximum values.

Patient characteristics and other baseline data (demographics, disease characteristics) will be summarized.

All data analyses will be performed using the SAS version 9.4 statistical software

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years at the day of consenting;
* Histologically confirmed diagnosis of Soft Tissue Sarcoma (STS) excepted GIST.
* Metastatic disease or unresectable locally advanced malignancy for which standard therapy by anthracycline is decided;
* At least one measurable lesion as per RECIST version 1.1.;
* ECOG Performance Status of 0-2;
* Patients must have an adequate organ and bone marrow function at baseline;
* Patient should understand, sign, and date the written voluntary informed consent form prior to any protocol-specific procedures performed and should be able and willing to comply with procedures as per protocol;
* Covered by a medical insurance.

Exclusion Criteria:

* Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results;
* Prior treatment with anthracycline;
* History of other malignancy other than study disease (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix) unless the patient has been free of disease for at least 3 years;
* Metabolic syndrome;
* Pregnant or breast-feeding woman criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
To develop a method for detecting and sorting CTCs (circulating tumour cells) from liquid biopsies (fresh blood samples) in patients with advanced or metastatic soft tissue sarcomas | 48 months
  Percentage of patients with detectable CTC

SECONDARY OUTCOMES:
Characterise the genetic profile of CTCs | 48 months
  Transcriptomic data Genomic data Percentage of organoids formed Changes in CTC counts
Establish tumour organoids from CTCs harvested before any initial treatment and, where possible, at the time of the first tumour recurrence | 48 months
  Transcriptomic data Genomic data Percentage of organoids formed Changes in CTC counts
Correlate the clinical response to treatments with the in vitro efficacy of the same treatments on tumour organoids. | 48 months
  progression free survival according RECIST 1.1 criteria
Assess the role of CTCs in tumour monitoring | 48 months
  progression free survival according RECIST 1.1 criteria
Evaluate the mechanisms of resistance to chemotherapy | 48 months
  progression free survival according RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- BRAHMI Mehdi, Lyon, France